CLINICAL TRIAL: NCT02845700
Title: Perceptual Retraining to Reduce Suicide Risk
Acronym: PRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Southeast Louisiana Veterans Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Wen Li, Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A-16054.13a
Record Dates: First submitted 2016-07-06; First posted 2016-07-27 (Estimated); Results first posted 2019-01-14 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2017-08

CONDITIONS: Perceptual Olfactory Bias

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Perceptual Retraining Treatment (PRT) (Active Comparator): The Perceptual Retraining Treatment will involve systematic presentation of diluted malodors. For each individual, vials on either side of their initial ideographic detection threshold will be presented. During the retraining, participants will be given feedback to shift their bias away from the malodorous target stimuli. For example, in the context of diluted solutions participants will be given the feedback that they are "correct" when a "neutral" response is given to solutions that are above the starting threshold (stronger malodor) and "incorrect" when a target is endorsed that is below the starting threshold (weaker malodor). Each training session will consist of 4 training blocks.
  Interventions: Behavioral: Perceptual Retraining Treatment
- Sham Neutral Training (SNT) (Placebo Comparator): Approximately half of the participants will be randomized to the SNT condition designed to control for the effects of time and learning. In the SNT condition, participants will complete the same assessments (including the olfactory bias assessment), as well as a sham training consisting of neutral/neutral odor pairing dilutions, rather than the combat/neutral odor pairings as in the PRT. Following the one-month assessment, they will be given the option to complete the PRT.
  Interventions: Behavioral: Sham Neutral training

INTERVENTIONS:
Behavioral: Perceptual Retraining Treatment — Perceptual retraining involves the systematic presentation of diluted malodors (i.e., odors perceived as threatening). For each individual, vials on either side of a pre-determined and ideographic detection threshold will be presented. During the retraining, participants will be given feedback to shift their bias away from the malodorous target stimuli. For example, in the context of diluted solutions participants will be given the feedback that they are "correct" when a "neutral" response is given to solutions that are above the starting threshold (stronger malodor) and "incorrect" when a target is endorsed that is below the starting threshold (weaker malodor).
  Arms: Perceptual Retraining Treatment (PRT)
Behavioral: Sham Neutral training — Control condition using systematic presentation of diluted neutral-neutral odor pairs.
  Arms: Sham Neutral Training (SNT)

SUMMARY:
The study will use a prospective design consisting of three phases. The phases are:

1. the development of the perceptual retraining treatment (PRT),
2. the evaluation of the treatment's feasibility and acceptability, and
3. an assessment of its efficacy.

During the third phase, a pilot study will be conducted in which participants will be randomly assigned to either PRT or a waitlist control group in order to assess efficacy. Diagnostic information and eligibility criteria will be assessed using the Structured Clinical Interview for Diagnostic and Statistical Manual (DSM) 4th ed. (SCID) and the Clinician Administered PTSD Scale for DSM-5 (CAPS-5).

DETAILED DESCRIPTION:
This study will use clinical interviews, self-report measures, and behavioral assessments to evaluate the efficacy of the PRT protocol. The study will recruit approximately 30 veterans. The primary inclusionary criterion will be that participants must show some evidence of olfactory perceptual bias toward military-relevant stimuli (e.g., burning rubber, decay, fuel). Investigators are not requiring current suicidal ideation as an entry criterion because investigators believe that a fair percentage of veterans will have some suicidal ideation/intent but making this an entry requirement will limit the investigators ability to recruit given the tight timeline for the study.

The study will consist of the development and evaluation of a novel intervention. The essential feature of this intervention is the use of a gradient of triggering smells (e.g., burning rubber, decay, fuel, etc.), to which participants will be systematically exposed in an effort to facilitate habituation to these odors. The PRT protocol will be administered over two 1-hour sessions. Participants will return 1 month after their final PRT protocol session to complete a battery of follow-up measures, as well as the CAPS-5.

The primary outcome measures of interest are: olfactory perceptual bias (as measured by the olfactory bias assessment), suicidal ideation and behaviors (as measured by the Beck Suicide Scale and Depressive Symptom Inventory- Suicidality Subscale), and symptoms related to suicide, such as anxiety and trauma (as measured by the Beck Anxiety Inventory and PTSD Checklist for DSM-5, respectively).

ELIGIBILITY:
Inclusion Criteria:

* evidence of olfactory perceptual bias toward military-relevant stimuli (e.g., burning rubber, decay, fuel).
* military combat exposure in Operation Iraqi Freedom, Enduring Freedom, or New Dawn.
* Age 18-60.

Exclusion Criteria:

* Significant medical illness that compromises olfactory perception or tolerance (e.g., significant olfactory disease or dysfunction, cardiovascular disease, respiratory disorders, renal disease, epilepsy, stroke, and uncontrolled hypertension or migraines).
* Evidence of imminent suicidal intent
* Evidence of current or past psychotic-spectrum disorders, or uncontrolled bipolar disorder.
* English speakers.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2015-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wen Li, PhD, Principal Investigator — Florida State University; Laurel Franklin, PhD, Principal Investigator — Southeastern Louisiana Veterans Health Care System
Locations (2):
- United States (2):
  - Florida State University, Tallahassee, Florida
  - Southeast Louisiana Veterans Health Care System, New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the community. Assessments occurred at the Florida State University Anxiety and Behavioral Health Clinic. In total, 16 individuals were assessed for eligibility. Of these, 15 participants were randomized to an intervention condition, and 1 was excluded because they were not combat exposed.
Pre-assignment Details: Of the 15 participants randomized to condition, 2 did not receive their allocated intervention (both in the Sensory Retraining Treatment [i.e., active] condition), because they withdrew from the study before the baseline appointment.
Groups:
- Perceptual Retraining Treatment (PRT): The retraining portion (PRT) will also involve the systematic presentation of diluted malodors. For each individual, vials on either side of their initial ideographic detection threshold established in the bias assessment phase will be presented. Participants will be given feedback to shift their bias away from the malodorous target stimuli. In the context of diluted solutions participants will be given the feedback that they are "correct" when a "neutral" response is given to solutions that are above the starting threshold (stronger malodor) and "incorrect" when a target is endorsed that is below the starting threshold (weaker malodor).
- Sham Neutral Training (SNT): Approximately half of the participants will be randomized to the Sham Neutral Training (SNT) ondition designed to control for the effects of time and learning. In the SNT condition, participants will complete the same assessments (including the olfactory bias assessment), as well as a sham training consisting of neutral/neutral odor pairing dilutions, rather than the combat/neutral odor pairings as in the PRT. Following the one-month assessment, they will be given the option to complete the PRT.
Period: Baseline Appointment
Arm/Group | Perceptual Retraining Treatment (PRT) | Sham Neutral Training (SNT)
Started | 6 | 7
Completed | 6 | 7
Not Completed | 0 | 0
Period: Intervention Session 1
Arm/Group | Perceptual Retraining Treatment (PRT) | Sham Neutral Training (SNT)
Started | 5 (1 participant withdrew after completing the Baseline Appointment) | 6 (1 participant withdrew after completing the Baseline Appointment)
Completed | 5 | 6
Not Completed | 0 | 0
Period: Intervention Session 2
Arm/Group | Perceptual Retraining Treatment (PRT) | Sham Neutral Training (SNT)
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0
Period: Month 1 Follow-Up
Arm/Group | Perceptual Retraining Treatment (PRT) | Sham Neutral Training (SNT)
Started | 2 (3 participants withdrew after completing the Intervention 2 Appointment) | 4 (2 participants withdrew after completing the Intervention 2 Appointment)
Completed | 2 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sensory Retraining Treatment (SRT): The retraining portion (SRT) will also involve the systematic presentation of diluted malodors. For each individual, vials on either side of their initial ideographic detection threshold established in the bias assessment phase will be presented. During the retraining, participants will be given feedback to shift their bias away from the malodorous target stimuli. For example, in the context of diluted solutions participants will be given the feedback that they are "correct" when a "neutral" response is given to solutions that are above the starting threshold (stronger malodor) and "incorrect" when a target is endorsed that is below the starting threshold (weaker malodor).
- Sham Neutral Training (SNT): Approximately half of the participants will be randomized to the SNT condition designed to control for the effects of time and learning. In the SNT condition, participants will complete the same assessments (including the olfactory bias assessment), as well as a sham training consisting of neutral/neutral odor pairing dilutions, rather than the combat/neutral odor pairings as in the SRT. Following the one-month assessment, they will be given the option to complete the SRT.
- Total: Total of all reporting groups
Arm/Group | Sensory Retraining Treatment (SRT) | Sham Neutral Training (SNT) | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.33 (13.63) | 32.71 (6.21) | 34.85 (10.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 7 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 7 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 4 | 2 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Olfactory Perceptual Bias
Description: A participant's ability to detect an array of threatening malodor in neutral dilution gradients will be tested at baseline and after the second and final intervention session (one week after baseline). Perceptual bias is calculated as the percentage of correct responses (i.e., yes or no to detecting the malodor) on an odor over 6 trials for each of the 8 odors, at 25% and 33% dilution (i.e., over 96 trials). Larger positive percentages indicate greater habituation to the malodor, and therefore a training effect toward reducing threat bias (i.e., a positive effect on intervention outcomes).
Time Frame: Baseline, Week 1
Measure: Mean (Standard Deviation); unit: Percent of correctly identified odors
Arm/Group | Perceptual Retraining Treatment (PRT) | Sham Neutral Training (SNT)
Number analyzed (Participants) | 5 | 6
Percent of correctly identified odors | 21.33 (25.67) | -5 (23.7)
Statistical Analysis 1: Comparison: Perceptual Retraining Treatment (PRT) vs Sham Neutral Training (SNT); Test type: Superiority; p = .08, ANOVA; 2 (time) x 2 (group) x 5 (dilution %) repeated measures ANOVA

2. Secondary Outcome: Change From Baseline in Mean Clinician Administered PTSD Scale for DSM-5 (CAPS-5) at 1 Month
Description: The Clinician Administered PTSD Scale for Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 (CAPS-5) was administered at the baseline appointment and 1-month follow-up appointment to assess PTSD symptom severity. All 20 of the CAPS-5 items are scored 0-4 and summed to calculate a total score, which ranges from 0-80. Higher scores indicate greater PTSD symptom severity. A difference score was calculated by subtracting the CAPS-5 score at 1-month from baseline, and averaged across each condition; thus, higher (positive) change scores are indicative of increases in PTSD symptom severity, whereas lower (negative) change scores are indicative of decreases in PTSD symptom severity.
Time Frame: Baseline, month 1
Measure: Mean (Standard Deviation); unit: Score on the CAPS-5
Arm/Group | Perceptual Retraining Treatment (PRT) | Sham Neutral Training (SNT)
Number analyzed (Participants) | 2 | 3
Score on the CAPS-5 | -16.00 (19.80) | 2.00 (16.71)
Statistical Analysis 1: Comparison: Perceptual Retraining Treatment (PRT) vs Sham Neutral Training (SNT); Post-hoc estimates of observed power for the difference between group means was calculated to be .15; Test type: Superiority; p = .39, t-test, 2 sided; t(4) = -1.19, p = .39

3. Secondary Outcome: Change in Suicidal Ideation Assessed Using the Depressive Symptom Inventory - Suicidality Subscale
Description: The Depressive Symptom Inventory - Suicidality Subscale (DSI-SS) was administered at the baseline appointment and 1 month follow-up appointment to assess the severity of thoughts related suicidal ideation. All four items of the DSI-SS are scored on a 0-3 scale, with total possible sum scores ranging from 0-12; higher scores indicate greater severity of suicidal ideation. For the outcome measure reported, a difference score was calculated by subtracting DSI-SS scores at 1 month from DSI-SS scores at baseline, and averaged across conditions. DSI-SS change scores of zero reflect no change from baseline to 1 month.
Time Frame: Baseline, month 1
Measure: Mean (Standard Deviation); unit: Scores on the DSI-SS
Arm/Group | Perceptual Retraining Treatment (PRT) | Sham Neutral Training (SNT)
Number analyzed (Participants) | 2 | 4
Scores on the DSI-SS | 0 (0) | 0 (0)

4. Secondary Outcome: Change in Beck Suicide Scale Scores From Baseline to 1 Month
Description: The Beck Suicide Scale (BSS) was administered at the baseline appointment and 1-month follow-up appointment to assess thoughts and behaviors related to suicidal ideation, desire, and attempts. The BSS comprises 21 items rated on a 0-3 scale. The first 19 items are sum scored with total possible scores ranging from 0 - 38, with higher scores indicating greater severity of suicide risk. A difference scores was calculated by subtracting the BSS score at 1 month from BSS scores at baseline. Mean change scores of 0 reflect no change in BSS scores from baseline to 1 month.
Time Frame: Baseline, month 1
Measure: Mean (Standard Deviation); unit: Scores on the BSS
Arm/Group | Perceptual Retraining Treatment (PRT) | Sham Neutral Training (SNT)
Number analyzed (Participants) | 2 | 4
Scores on the BSS | 0 (0) | 0 (0)

5. Secondary Outcome: Change in the Beck Anxiety Inventory-II From Baseline to 1 Month
Description: The Beck Anxiety Inventory-II (BAI) was administered at the baseline appointment and 1-month follow-up appointment to assess symptom severity associated with anxious arousal. The BAI comprises 21 items rated on a 0-3 scale, which can be sum scored to calculate total scores ranging from 0 - 63. Higher scores on the BAI are indicative of greater anxious arousal. A difference scores was calculated by subtracting the BAI score at 1 month from BAI scores at baseline; thus, higher (positive) change scores are indicative of increases in anxious arousal, whereas lower (negative) change scores are indicative of decreases in anxious arousal.
Time Frame: Baseline, month 1
Measure: Mean (Standard Deviation); unit: Scores on the BAI
Arm/Group | Perceptual Retraining Treatment (PRT) | Sham Neutral Training (SNT)
Number analyzed (Participants) | 2 | 4
Scores on the BAI | -3.50 (.71) | -1.75 (3.5)
Statistical Analysis 1: Comparison: Perceptual Retraining Treatment (PRT) vs Sham Neutral Training (SNT); Post-hoc estimates of observed power for the difference between group means was calculated to be .08; Test type: Superiority; p = .54, t-test, 2 sided; t(4) = 0.66, p = .54

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Sensory Retraining Treatment (SRT) | Sham Neutral Training (SNT)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 0/6 | 0/7

LIMITATIONS AND CAVEATS:
Overall sample size was limited due to delays of project approval at the Southeast Louisiana Veterans Health Care System site. Early terminations at the Florida State University site further lead to small numbers of subjects to be analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No